CLINICAL TRIAL: NCT04629144
Title: Multicenter Randomized Double-blind Study Comparing the Efficacy and Safety of Belimumab in the Treatment of Non-infectious Active Cryoglobulinemia Vasculitis Compared to Placebo. TRIBECA STUDY (Treatment nd BElimumab in Cryoglobulinemia Associated Vasculitis)
Brief Title: Efficacy and Safety of Belimumab in the Treatment of Non-infectious Active Cryoglobulinemia Vasculitis Compared to Placebo. TRIBECA STUDY (Treatment nd BElimumab in Cryoglobulinemia Associated Vasculitis)
Acronym: TRIBECA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APHP180351
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Vasculitis; Cryoglobulinemia
Keywords: Belimumab; Vasculitis; Cryoglobulinemia; Non-infectious
MeSH Terms: conditions — Vasculitis; Cryoglobulinemia | interventions — belimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Belimumab (Experimental): Belimumab administered subcutaneously 200mg weekly from week 1 to week 24.
  Interventions: Drug: Belimumab
- Placebo (Placebo Comparator): Placebo of Belimumab administered subcutaneously weekly from week 1 to week 24.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belimumab — Belimumab administered subcutaneously 200mg weekly from week 1 to week 24.
  Both arms will have the same corticosteroid tapering scheme, with an initial dose of 30 mg/day. The following schedule of reduction of prednisone will apply to both groups as long as the disease is inactive:
  * 30 mg/day week (W)0-W2,
  * 20 mg/day W2-W4
  * 15 mg/day W4-W6,
  * 10 mg/day W6-W8,
  * 5 mg/day W8-W10
  Between W10-W12 the strategy for stopping glucocorticoids is left to the investigator's discretion.
  Stopping glucocorticoid therapy at W12. At each step, the prednisone dose will be reduced only in the absence of signs of vasculitis activity.
  Arms: Belimumab
Drug: Placebo — Both arms will have the same corticosteroid tapering scheme, with an initial dose of 30 mg/day. The following schedule of reduction of prednisone will apply to both groups as long as the disease is inactive:
  * 30 mg/day week (W)0-W2,
  * 20 mg/day W2-W4
  * 15 mg/day W4-W6,
  * 10 mg/day W6-W8,
  * 5 mg/day W8-W10
  Between W10-W12 the strategy for stopping glucocorticoids is left to the investigator's discretion.
  Stopping glucocorticoid therapy at W12. At each step, the prednisone dose will be reduced only in the absence of signs of vasculitis activity.
  Arms: Placebo

SUMMARY:
Cryoglobulinemia vasculitis (CV) is a systemic immune-mediated small vessel vasculitis. Rituximab proved effective on main vasculitis signs, with a complete clinical response of 65%. However, CV relapse is noted in up to 40% of patients. Following rituximab, serum Blys concentration significantly increased and may favor relapses. Tribeca is a multicentre randomized controled study comparing safety and efficacy of belimumab to placebo in non infectious cryoglobulinemia vasculitis.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria will be checked at the inclusion/randomization visit. Patients meeting the following criteria may be included in the study:

1. Age > 18 years
2. Written inform consent
3. Active mixed cryoglobulinemia vasculitis, at initiation of rituximab, define by a. a clinically active vasculitis with skin, joint, renal, peripheral nerve, central neurological, digestive, pulmonary and/or cardiac involvement , b. history of positive cryoglobulinemia and/or positive Rheumatoid factor associated with low C4 complement level , and/or a monoclonal component (IgM Kappa) and/or a histologal proof of vasculitis in the affected organs
4. Affiliated to National French social security system
5. Having received Rituximab as induction therapy within 6 weeks (1 to 4 infusions, dose at the discretion of the investigator)
6. Female subjects of childbearing potential must have a negative serum or urinary pregnancy test at inclusion visit, and confirmed monthly while in study, out to at least 92 days (5 half lives) post last dose.
7. For subjects with reproductive potential (male or female), a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study from 2 weeks prior to administration of the 1st dose of study agent until 92 days after the last dose of study agent. Therefore the subjects agree to 1 of the following:

   1. Complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 92 days after the last dose of study agent (Sexual inactivity by abstinence must be consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception) OR
   2. Consistent and correct use of 1 of the following acceptable methods of birth control for 1 month prior to the start of the study agent, during the study, and 92 days after the last dose of study agent o Oral contraceptive, either combined or progestogen alone o Injectable progestogen o Implants of levonorgestrel or etonogestrel o Estrogenic vaginal ring o Percutaneous contraceptive patches o Intrauterine device (IUD) or intrauterine system (IUS) with <1% failure rate as stated in the product label

      o Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records
      * Double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository) These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring subjects understand how to properly use these methods of contraception.
8. HIV negative serology ; negative HBs Ag test and HBc Ab test; HCV negative serology or negative HCV RNA if positive HCV serology within 3 months before inclusion:

   o In case of negative AgHBs and positive HBc Ab test, HBV DNA test must be negative; AND Hepatitis B surveillance should be started (monthly HBsAg and HBV DNA testing for the duration of the study treatment and at least every 12 weeks after treatment is discontinued for the duration of study treatment. In addition, antiviral prophylaxis should be started before the first administration of the study treatment and continued until 12 months after completion of study treatment; HCV negative serology or negative HCV RNA if positive HCV serology within 3 months before inclusion
9. neutrophils (ANC) >1x109/L

Exclusion criteria :

Subjects will be not included from the study if they meet any of the following criteria:

1. Patient with a vasculitis unrelated to cryoglobulinemia
2. Patient with non active cryoglobulinemia vasculitis, at initiation of rituximab. Patients with mixed inactive vasculitis following rituximab administration may be included.
3. Excluded concomitant medications:

   1. 365 days Prior to Investigational Medicinal Product (Belimumab or placebo):: Any biologic investigational agent (e.g., abetimus sodium, anti CD40L antibody, BG9588/ IDEC 131) Investigational agent applies to any drug not approved for sale in the country in which it is being used
   2. 180 Days Prior to Investigational Medicinal Product (Belimumab or placebo):: Intravenous cyclophosphamide
   3. 30 Days Prior to Investigational Medicinal Product (Belimumab or placebo): (or 5 half lives, whichever is greater) Any non-biologic investigational agent Investigational agent applies to any drug not approved for sale in the country in which it is being use
   4. Live vaccines within 30 days prior to baseline or concurrently with Investigational Medicinal Product (Belimumab or placebo)
4. Have a history of malignant neoplasm within the last 5 years, other than carcinoma in situ of the cervix or excised basal cell, squamous cell carcinoma of the skin and low grade hemopathy with no indication for a specific treatment
5. Have evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, pose a significant suicide risk
6. Have a Progressive multifocal leukoencephalopathy
7. Have a history of a primary immunodeficiency

9. Have a history of major organ transplant or hematopoietic stem cell/marrow transplant or renal transplant

10. Infection history:

* Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus
* Infection requiring hospitalization and/or use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti-parasitic agents) within 60 days of the inclusion visit.

  11. Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to the inclusion visit

  12. Have a historically positive HIV test according to results obtained within 3 months prior to inclusion visit

  13. Hepatitis status according to results obtained within 3 month prior to inclusion visit :
* Positive test for hepatitis B RNA
* Positive test for Hepatitis C RNA

  14. Have a history of a hypersensitivity or an anaphylactic reaction to parenteral administration of Belimumab, corticosteroids or any excipients of the treatments administered during the study

  15. If Women of Child Bearing Potential (WCBP) are included please see special instructions in Inclusion criteria

  16. Pregnant or breast feeding women

  17. Have any intercurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study

  18. Patients under legal protection or unable to consent

  19. Participation to another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Complete clinical response rate at week 25 with corticosteroid withdrawal at week 12 | Week 25
  Complete clinical response is defined by remission of all affected organs involved at baseline and the absence of clinical relapse.
  * Skin and articular remissions
  * Renal remission
  * Neurological remission
  * Digestive remission
  * Cardiac remission
  * Central nervous system remission
  * Pulmonary remission

SECONDARY OUTCOMES:
Safety W25 | Week 25
  Frequency and severity of adverse clinical events
Safety W48 | Week 48
  Frequency and severity of adverse clinical events
Response W13 | Week 13
  The complete clinical response is defined by the remission of all affected organs involved at baseline and the absence of clinical relapse.
  Partial clinical response The partial clinical response is defined by the improvement and / or remission of more than half of the organ involvement present at baseline and the absence of clinical relapse.
  No clinical response Patients with no clinical response at W4 will be defined by worsening of ulcers or cutaneous necrosis, worsening peripheral neurological involvement or by persistence of active renal involvement defined by persistence of proteinuria> 1.5 g / 24h or proteinuria/creatinuria <150 mg/mmol).
Response W25 | Week 25
  The complete clinical response is defined by the remission of all affected organs involved at baseline and the absence of clinical relapse.
  Partial clinical response The partial clinical response is defined by the improvement and / or remission of more than half of the organ involvement present at baseline and the absence of clinical relapse.
  No clinical response Patients with no clinical response at W4 will be defined by worsening of ulcers or cutaneous necrosis, worsening peripheral neurological involvement or by persistence of active renal involvement defined by persistence of proteinuria> 1.5 g / 24h or proteinuria/creatinuria <150 mg/mmol).
Response W48 | Week 48
  The complete clinical response is defined by the remission of all affected organs involved at baseline and the absence of clinical relapse.
  Partial clinical response The partial clinical response is defined by the improvement and / or remission of more than half of the organ involvement present at baseline and the absence of clinical relapse.
  No clinical response Patients with no clinical response at W4 will be defined by worsening of ulcers or cutaneous necrosis, worsening peripheral neurological involvement or by persistence of active renal involvement defined by persistence of proteinuria> 1.5 g / 24h or proteinuria/creatinuria <150 mg/mmol).
Rate of cryoglobulinemia clearance W13 | Week 13
  cryoglobulinemia clearance
Rate of cryoglobulinemia clearance W25 | Week 25
  cryoglobulinemia clearance
Rate of cryoglobulinemia clearance W48 | Week 48
  cryoglobulinemia clearance
rheumatoid factor activity W13 | Week 13
  negativation of rheumatoid factor activity
rheumatoid factor activity W25 | Week 25
  negativation of rheumatoid factor activity
rheumatoid factor activity W48 | Week 48
  negativation of rheumatoid factor activity
C4 complement level W13 | Week 13
  normalization of C4 complement level
C4 complement level W25 | Week 25
  normalization of C4 complement level
C4 complement level W48 | Week 48
  normalization of C4 complement level
Early failures | Week 5
  Rate of early failures (non clinical response at W5) Patients with no clinical response at W4 will be defined by worsening of ulcers or cutaneous necrosis, worsening peripheral neurological involvement or by persistence of active renal involvement defined by persistence of proteinuria> 1.5 g / 24h or proteinuria/creatinuria <150 mg/mmol,).
Clinical relapse rate W48 | Week 48
  Relapse is defined as de novo appearance or recurrence of a manifestation of cryoglobulinemia vasculitis
Prednisone W25 | Week 25
  Cumulative dose of prednisone
Prednisone W48 | Week 48
  Cumulative dose of prednisone
Gammaglobulin | Baseline
Gammaglobulin | Week 48
CD19+ | Baseline
CD19+ | Week 48
Quality of life W25 | Week 25
  Quality of life score SF-36. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software for the commercial version, but no special software is needed for the RAND-36 version. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health
Quality of life W48 | Week 48
  Quality of life score SF-36. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. To calculate the scores it is necessary to purchase special software for the commercial version, but no special software is needed for the RAND-36 version. Pricing depends on the number of scores that the researcher needs to calculate.
  The eight sections are:
  vitality physical functioning bodily pain general health perceptions physical role functioning emotional role functioning social role functioning mental health
Infections | Week 48
  Rate of infections
BVAS activity W13 | Week 13
  BVAS activity score as defined in Flossmann, Oliver, et al. "Development of comprehensive disease assessment in systemic vasculitis." Postgraduate medical journal 84.989 (2008): 143-152.
BVAS activity W25 | Week 25
  BVAS activity score as defined in Flossmann, Oliver, et al. "Development of comprehensive disease assessment in systemic vasculitis." Postgraduate medical journal 84.989 (2008): 143-152.
BVAS activity W48 | Week 48
  BVAS activity score as defined in Flossmann, Oliver, et al. "Development of comprehensive disease assessment in systemic vasculitis." Postgraduate medical journal 84.989 (2008): 143-152.

OTHER OUTCOMES:
Immunomonitoring W13 | Week 13
  deep immunophenotyping, cytokines production, clonal IgM memoryCD21-/low cells) description
Immunomonitoring W25 | Week 25
  deep immunophenotyping, cytokines production, clonal IgM memoryCD21-/low cells) description
Immunomonitoring W48 | Week 48
  deep immunophenotyping, cytokines production, clonal IgM memoryCD21-/low cells) description
renal response W13 | Week 13
  Renal remission is evaluated biologically (proteinuria <0.5g/24h or proteinuria/creatinuria <50 mg/mmol).
renal response W25 | Week 25
  Renal remission is evaluated biologically (proteinuria <0.5g/24h or proteinuria/creatinuria <50 mg/mmol).

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - CH Blois, Blois
  - CHU (Haut-Lévêque), Bordeaux
  - CHU Caen, Caen
  - Hopital Henri Mondor, Créteil
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - CHU La Conception, Marseille
  - CHU Nantes, Nantes
  - CH Nimes, Nîmes
  - Hopital de La Pitié Salpetriere AP-HP, Paris
  - Hopital Européen Georges Pompidou, Paris
  - Hopital Necker, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Hopital Tenon, Paris
  - CHU Starsbourg, Strasbourg
  - Hopital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CHU Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided